CLINICAL TRIAL: NCT02554851
Title: Efficacy and Safety Evaluation of the Intralesional Recombinant Human Epidermal Growth Factor (rhEGF) in Subjects With Diabetic Foot Ulcer. Multicenter, Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Efficacy and Safety Evaluation of the Intralesional Recombinant Human Epidermal Growth Factor (rhEGF) in Subjects With Diabetic Foot Ulcer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASCLIN002/2015
Record Dates: First submitted 2015-09-11; First posted 2015-09-18 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Foot Ulcer, Diabetic; Epidermal Growth Factor
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): This group will receive the standard medication and the placebo drug
  Interventions: Other: Placebo
- recombinant human Epidermal Growth Fact (Experimental): This group will receive the standard medication and the recombinant human Epidermal Growth Factor (HEBERPROT)
  Interventions: Drug: recombinant human Epidermal Growth Factor (rhEGF)

INTERVENTIONS:
Drug: recombinant human Epidermal Growth Factor (rhEGF) — The Heberprot-P® is a parenteral formulation, which is in a lyophilized powder vial presentation containing 75μg of recombinant Epidermal Growth Factor (rhEGF) for local application (intralesional) with the therapeutic potential to promote granulation and wound healing of DFU. The rhEGF is a polypeptide of 53 amino acids and has the ability to stimulate fibroblasts, keratinocytes and vascular endothelial cells proliferation. Then it contributes to its properties in scar tissue formation. The action mechanism is based on the interaction with specific receptors located on specifics cell membranes. The rhEGF was developed through recombinant DNA technology and it has been produced by biotechnological methods in Saccharomyces cerevisiae yeast line.
  Other Names: Heberprot-P®
  Arms: recombinant human Epidermal Growth Fact
Other: Placebo — This group will receive the standard medication and the placebo drug. The placebo drug has the same formulation, except for the fact that it does not contain the recombinant human Epidermal Growth Factor (rhEGF).
  Arms: placebo

SUMMARY:
Phase III clinical trial, multicenter, controlled, randomized, double-blind, with two parallel groups (experimental and control). Both study groups will receive standard therapy currently available in treatment centers for diabetic foot ulcer (DFU). Associate with the standard therapy, it will be given the recombinant human Epidermal Growth Factor (rhEGF) to experimental group and in the control group, it will be given a formulation without pharmacological effect (placebo) in order to masking and control of intralesional application. Participants with type 1 and type 2 diabetes mellitus (DM) diagnosed with DFU for at least 4 weeks, treated in referral centers participating in the study, agreeing to participate after reading, understanding and signing of Informed Consent (IC); meet all the inclusion criteria; and presenting no exclusion criteria. The Informed Consent (IC) should be applied to potential participants, as recommended by the regulations and ethical consensus before beginning any procedure related to the clinical trial. In the early weeks, participants will be evaluated at the research centers by the study team (doctors and / or staff). The number of visits will be determined by the investigator, thus ensuring appropriate assistance to participants, and avoiding any complications with DFU. By meeting the eligibility requirements (inclusion and exclusion criteria), the participant will undergo a thorough evaluation of the DFU before the start of treatment. This assessment is precisely to classify the condition of the ulcer before treatment and provide relevant information for statistical analysis of the protocol. If eligible, the participant will be randomly set to treatment arm (placebo or rhEGF) and the administration of investigational product associated with predefined standardized outpatient therapy will be initiated. This administration occurs three times per week until the DFU is scarred, not exceeding 8 weeks of treatment (T.01 to T.08) .The study will be randomized and balanced according to the type and size of the DFU. This balancing is necessary to ensure that both treatment groups are homogeneous for participants under different conditions. All participants will be applied established standard therapy for the treatment of DFU. The objective is to provide regular care for healing and reduce possible bias in the efficacy analysis and product safety. After the treatment period (last dose of the experimental drug) the participant will start the follow-up period, with 16 weeks duration. The participant shall be subjected to weekly visits for ongoing assessment of DFU, however, according to the investigator, may result in unscheduled visits to assess local or general clinical events. After the monitoring period, the participant will be observed for 24 additional weeks, visits every 4 weeks (E.01 E.24 a) having beginning one week after the last visit of follow-up. This period is intended to assess possible events related to the efficacy and safety that can happen in the period, mainly for analysis of secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. DM type 1 or 2 diagnosis
2. DFU persisting for a minimum of 4 weeks If the participant have more than one DFU, then it will be treated the one with the largest extension and that follows the inclusion and exclusion criteria.
3. DFU 's rating according to the PEDIS system:Perfusion: grades 1 or 2; Extension: Area ≥ 2 cm2; Depth: grades 2 or 3; Infection: grades 1 or 2; Sensitivity: grade 2

If the consented participant is classified as having infection grade 3 without the presence of osteomyelitis, it will be possible to treat it with antibiotics empirically. However, randomization will be made only after this treatment and only if the infection has regressed to grade 1 or 2;

Exclusion Criteria:

1. Age less than 18 years;
2. Pregnancy or breastfeeding (women in childbearing age will need to use a contraception method);
3. Evidence of bone involvement : direct visualization of bone structures; positive survey (probe to bone) ; image investigation (simple x-ray or MRI);
4. Urgent or imminent need of amputation;
5. Eminent indication for revascularization;
6. Glycated hemoglobin (HbA1c) counted greater than 11 %
7. Use of drugs that can affect or contribute to the healing of ulcers as corticosteroids; immunosuppressive; chemotherapy; other growth factors;
8. Clinical signs of malnutrition or serum albumin <30 g / L;
9. Angina pectoris classified as 3 or 4 (according to the Canadian Cardiovascular Society Angina Classification);
10. Congestive heart failure class IV (according to the New York Heart Association);
11. Severe hepatic impairment, defined as ALT and / or AST greater than 5 (five) times the normal maximum reference value;
12. Acute renal failure, defined as serum creatinine levels equal or higher than 1.5 times the baseline value in the last 7 days (according to KDIGO and RIFLE classification);
13. End-stage renal disease (creatinine clearance equal or lower than 30 ml / min or on dialysis);
14. History or suspected neoplasia (according to previous laboratory tests, imaging or biopsy);
15. Psychiatric disorders that may alter the participants evaluation, or prevent proper consent and / or cognitive aspects that demonstrate the possibility of noncompliance with treatment or the adoption of aseptic criteria;
16. Occurrence of the following events 30 days prior to inclusion in the protocol: participation in other clinical studies; hypoglycemic coma (blood glucose less than or equal to 30 mg / dL with loss of consciousness or need for help); diabetic ketoacidosis or hyperosmolar state within 30 days prior to inclusion;
17. Occurrence of the following events 60 days prior to inclusion in the protocol: hospitalization for acute coronary syndrome, percutaneous intervention (eg cardiac, cerebrovascular, aortic) or greater cardiac surgery; myocardial infarction; cerebrovascular accident; cardiac arrest; sustained ventricular tachycardia; acute coronary syndrome, in investigator opinion; uncontrolled severe hypertension, defined as systolic blood pressure equal or higher than 180 mmHg and / or diastolic blood pressure equal or higher than 110 mmHg;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with 100% healing at the end of follow-up | up to 9 months
  Contingency tables for the proportion of participants with 100% healing at this time period (16th week of treatment evaluation) with their respective frequencies and percentages, according to the treatment group will be generated; 95% confidence intervals for the proportion of participants with 100% healing at the end of follow-up will be generated for each group; range of 95% confidence interval for the difference between the proportions of participants with 100% healing in each treatment group at the end of follow-up will be generated; the confirmatory data analysis will be held for proportions, one-sided, in order to verify the superiority hypothesis envisaged, the sample design.